CLINICAL TRIAL: NCT01478815
Title: Contingency Management for Persons With Severe Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-070-3; P30DA023918 (NIH)
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (Placebo Comparator)
  Interventions: Other: Standard Care
- Contingency management for abstinence from drugs (Experimental)
  Interventions: Behavioral: contingency management

INTERVENTIONS:
Behavioral: contingency management — Participants will receive the opportunity to win prizes for submitting cocaine negative urine samples.
  Arms: Contingency management for abstinence from drugs
Other: Standard Care — Standard Care
  Arms: Standard Care

SUMMARY:
Contingency management is efficacious for treating cocaine abuse, but contingency management interventions have rarely been applied to patients with severe and persistent mental health problems. This pilot project will estimate effect sizes of contingency management for reducing cocaine use in patients receiving psychiatric care at a large community based mental health program. In total, 30 cocaine abusing patients will be randomized to one of two 8-week treatment conditions: standard care or standard care with contingency management. Patients in both conditions will provide breath and urine samples for toxicology testing twice per week. In the contingency management condition, patients will receive the opportunity to win prizes for submitting cocaine negative urine samples. The investigators expect that patients receiving contingency management will evidence reductions in cocaine use and may show improvements in psychiatric symptoms and psychosocial functioning relative to patients in standard care. Effect size estimates obtained from this study will be used to guide larger scale and longer duration evaluations of contingency management for dually diagnosed patients.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* meet DSM-IV criteria for cocaine abuse or dependence
* English speaking
* pass a brief quiz regarding study procedures to ensure understanding of the informed consent process.

Exclusion Criteria:

* dementia
* in recovery from pathological gambling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
longest continuous period of cocaine abstinence | Week 8

SECONDARY OUTCOMES:
other drug use and psychosocial problems | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Petry, Ph.D., Principal Investigator — UConn Health
Locations (1):
- Community Mental Health Affiliates, Inc., New Britain, Connecticut, United States

REFERENCES:
- [Derived] Petry NM, Alessi SM, Rash CJ. A randomized study of contingency management in cocaine-dependent patients with severe and persistent mental health disorders. Drug Alcohol Depend. 2013 Jun 1;130(1-3):234-7. doi: 10.1016/j.drugalcdep.2012.10.017. Epub 2012 Nov 20. PMID 23182410